CLINICAL TRIAL: NCT02920060
Title: Levetiracetam Versus Sodium Valproate in Children With Refractory Generalized Convulsive Status Epilepticus : An Open Randomized Study
Brief Title: Levetiracetam Versus Sodium Valproate in Children With Refractory Generalized Convulsive Status Epilepticus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Collaborators: Institute of Medical Sciences of the Banaras Hindu University, India (Other)
Responsible Party: Principal Investigator, Dr. Astha Panghal, Pricipal investigator, Banaras Hindu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ECR/526/Inst/UP/2014
Record Dates: First submitted 2016-09-24; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Grand Mal Status Epilepticus
Keywords: RSE
MeSH Terms: conditions — Status Epilepticus | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental): patient in this group will receive intravenous levetiracetam as loading dose of 30 mg/kg at a rate of 50 mg/min
  Interventions: Drug: Intravenous levetiracetam
- Sodium valproate (Active Comparator): patients in this group will receive intravenous sodium valproate 20 mg/kg as loading dose at a rate of 40 mg/min
  Interventions: Drug: Sodium valproate

INTERVENTIONS:
Drug: Intravenous levetiracetam — intravenous levetiracetam(30mg/kg bolus followed by 20mg/kg/dose IV 12 hourly).
  Other Names: injection Levera
  Arms: Levetiracetam
Drug: Sodium valproate — intravenous sodium valproate(20mg/kg bolus followed by 10 mg/kg/dose IV 8hrly)
  Other Names: injection Encorate
  Arms: Sodium valproate

SUMMARY:
This study is a randomized, open label, parallel group,comparing the safety and efficacy of valproate and levetiracetam in patients of age group 1 to 16 years with status epilepticus not responded to phenytoin and benzodiazepines approaching to pediatric emergency , IMS, BHU. The primary outcome measures will be Proportion of children in either group who have Cessation of all clinical seizure within 30 min of drug administration and secondary outcome will be time taken to control seizure (minutes) from the initiation of infusion. Proportion of children in either group who required additional drugs to abort ongoing clinical seizures, rates of adverse events (hypotension, bradycardia, respiratory depression, PICU stay, in hospital mortality) in the two groups were measured. Refractory status epilepticus condition is major pediatric neurological emergency with high mortality and morbidity. Till now, the treatment guidelines for it are based primarily on retrospective studies with very few randomized studies. There is lack of sufficient data to recommend one drug over another for treatment of refractory status epilepticus.

DETAILED DESCRIPTION:
In our study patients were considered to have RSE if children were still having active convulsions despite receiving injection lorazepam intravenously at a dose of 0.1 mg/kg (max 4 mg) at a rate maximum upto 2 mg/min or intravenous diazepam at a dose of 0.2 - 0.3 mg/Kg (maximum 10 mg) slowly or intravenous midazolam at a dose of 0.15 - 0.2 mg/kg(max 5 mg). In case of children with difficult intravenous access buccal/nasal midazolam 0.2 - 0.3 mg/kg (maximum 5 mg) per rectal diazepam 0.5 mg/kg (maximum 10 mg) or intramuscular midazolam 0.2 mg/kg (maximum 5 mg). If seizure continued at 5 minutes, a repeat dose of benzodiazepine was given with same dose. At 10 minutes, if the seizure activity still remains intravenous phenytoin was given at a dose of 20mg/kg(maximum- 1000mg) at a rate of 1mg/kg/minute or intravenous fosphenytoin at 20mg PE/kg (if available) at a rate of 3mg PE/kg/minute.

Patients having seizure activity despite administration of above medications were considered to have RSE. Out of thousands of patients seen in outdoor and emergency ward, 80 patients were diagnosed to have RSE and met the inclusion criteria. After counselling the parents/guardians about the medications and obtaining a written informed consent they were randomized to into two groups : sodium valproate(V) and levetiracetam group(L), using a computer generated randomization chart. Forty patients in group V received intravenous valproic acid in dose of 20 mg/kg as loading dose at a rate of 40 mg/min after dilution with normal saline followed by maintenance dose of 10mg/kg/dose 8 hourly. In group L patients received intravenous levetiracetam as loading dose of 30 mg/kg at a rate of 50 mg/min followed by 20mg/kg/dose 12 hourly.

ELIGIBILITY:
Inclusion Criteria:

1. Age - 1 year to 16 years
2. Gender - male and female both
3. Refractory generalized convulsive status epilepticus i.e. not responding to any two of the first line drugs

Exclusion Criteria:

1. Patients with epilepsia partialis continua.
2. Patients with definite history of any allergic reaction to intravenous levetiracetam or intravenous valproate, or any contraindications in giving these drugs.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
cessation of convulsions (clinically evident motor activity) | 30 minutes
  clinical cessation of convulsions, vitals monitoring

SECONDARY OUTCOMES:
seizure activity at 24 hours of infusion | 24 hours
  whether clinical convulsive activity cessation or not
seizure recurrence | 24 hours
  average number of seizure recurring after drug infusion within 24 hours
additional number of drugs | 24 hours
  number of additional drugs to control RSE within 24 hours of infusion
time taken to control seizure activity | 24 hours
  time needed to control convulsive activity from infusion time
change in vital parameters after infusing interventional agent | 24 hours
  vital parameters will be recorded every 15 minutes for the first 1 hour after the intervention began and mean value of vital parameters will be compared in two groups
neurological outcome and seizure control | 1 month
  to look for any neurological deficit or behavioural abnormality and seizure control at one month of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rajniti Prasad, MD, Study Director — Banaras Hindu University

IPD SHARING:
Plan to Share IPD: No